CLINICAL TRIAL: NCT04804644
Title: Phase III Trial of Stereotactic Radiosurgery (SRS) Versus Hippocampal-Avoidant Whole Brain Radiotherapy (HA-WBRT) for Brain Metastases From Small Cell Lung Cancer
Brief Title: Testing if High Dose Radiation Only to the Sites of Brain Cancer Compared to Whole Brain Radiation That Avoids the Hippocampus is Better at Preventing Loss of Memory and Thinking Ability
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NRG-CC009; NCI-2020-11651 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-CC009 (Other: NRG Oncology); NRG-CC009 (Other: DCP); NRG-CC009 (Other: CTEP); UG1CA189867 (NIH)
Record Dates: First submitted 2021-03-09; First posted 2021-03-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Lung Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Brain; Recurrent Lung Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Small Cell Lung Carcinoma; Brain Neoplasms; Lung Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Memantine; Mental Status and Dementia Tests; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (SRS) (Experimental): Patients undergo SRS over 1 day (in some cases several days). Patients undergo blood sample collection and MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Neurocognitive Assessment; Radiation: Stereotactic Radiosurgery; Other: Survey Administration
- Arm II (HA-WBRT, memantine) (Active Comparator): Patients also undergo HA-WBRT QD for 2 weeks in the absence of disease progression or unacceptable toxicity. Patients will also receive memantine PO QD or BID for up to 24 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection and MRI throughout the study.
  Interventions: Procedure: Magnetic Resonance Imaging; Drug: Memantine Hydrochloride; Other: Neurocognitive Assessment; Other: Survey Administration; Radiation: Whole-Brain Radiotherapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm I (SRS)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Memantine Hydrochloride — Given PO
  Other Names: Ebixia; Namenda
  Arms: Arm II (HA-WBRT, memantine)
Other: Neurocognitive Assessment — Ancillary studies
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: SRS; Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
  Arms: Arm I (SRS)
Other: Survey Administration — Ancillary studies
Radiation: Whole-Brain Radiotherapy — Undergo HA-WBRT
  Other Names: WBRT; whole-brain radiation therapy
  Arms: Arm II (HA-WBRT, memantine)

SUMMARY:
This phase III trial compares the effect of stereotactic radiosurgery to standard of care memantine and whole brain radiation therapy that avoids the hippocampus (the memory zone of the brain) for the treatment of small cell lung cancer that has spread to the brain. Stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may cause less damage to normal tissue. Whole brain radiation therapy delivers a low dose of radiation to the entire brain including the normal brain tissue. Hippocampal avoidance during whole-brain radiation therapy (HA-WBRT) decreases the amount of radiation that is delivered to the hippocampus which is a brain structure that is important for memory. The drug, memantine, is also often given with whole brain radiotherapy because it may decrease the risk of side effects related to thinking and memory. Stereotactic radiosurgery may decrease side effects related to memory and thinking compared to standard of care HA-WBRT plus memantine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine whether stereotactic radiosurgery (SRS) relative to whole brain radiotherapy with hippocampal avoidance (HA-WBRT) plus memantine hydrochloride (memantine) for brain metastases from small cell lung cancer (SCLC) prevents cognitive function failure as measured by cognitive decline on a battery of tests: the Hopkins Verbal Learning Test - Revised (HVLT-R), Controlled Oral Word Association (COWA) test, and the Trail Making Test (TMT).

SECONDARY OBJECTIVES:

I. Determine whether SRS relative to HA-WBRT plus memantine for brain metastases from SCLC preserves cognitive function as separately measured by the HVLT-R, COWA, TMT Parts A and B, and Clinical Trial Battery Composite (CTB COMP).

II. Assess perceived difficulties in cognitive abilities using Patient Reported Outcomes Measurement Information System (PROMIS) after SRS relative to HA-WBRT plus memantine for brain metastases from SCLC.

III. Assess symptom burden using the MD Anderson Symptom Inventory for brain tumor (MDASI-BT) after SRS relative to HA-WBRT plus memantine for brain metastases from SCLC.

IV. Compare cumulative incidence of intracranial disease progression after SRS relative to HA-WBRT plus memantine for brain metastases from SCLC.

V. Compare overall survival after SRS relative to HA-WBRT plus memantine for brain metastases from SCLC.

VI. Compare cumulative incidence of neurologic death after SRS relative to HA-WBRT plus memantine for brain metastases from SCLC.

VII. Compare the number of salvage procedures used to manage recurrent intracranial disease following SRS relative to HA-WBRT plus memantine for SCLC brain metastases.

VIII. Compare adverse events between the treatment arms according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 criteria.

IX. Compare the risk of developing cerebral necrosis between SRS and HA-WBRT plus memantine in patients receiving concurrent immunotherapy.

EXPLORATORY OBJECTIVES:

I. Compare cumulative incidence of local brain recurrence, distant brain relapse, and leptomeningeal dissemination after SRS relative to HA-WBRT plus memantine for brain metastases from SCLC.

II. Compare the cost of brain-related therapies and quality-adjusted life years in patients who receive SRS relative to HA-WBRT plus memantine for brain metastases from SCLC.

III. Evaluate the time delay to salvage WBRT or HA-WBRT in patients enrolled on the SRS arm.

IV. Evaluate whether a time delay for chemotherapy has an effect on overall survival in patients receiving HA WBRT plus memantine relative to SRS for brain metastases from SCLC.

V. Evaluate baseline magnetic resonance (MR) imaging biomarkers of white matter injury and hippocampal volumetry as potential predictors of cognitive decline and differential benefit from SRS relative to HA-WBRT plus memantine for brain metastases from SCLC.

VI. Evaluate the correlation between neurocognitive functioning and patient-reported outcomes.

VII. Collect serum, plasma and imaging studies for future translational research analyses.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo SRS over 1 day (in some cases several days).

ARM II: Patients undergo HA-WBRT once daily (QD) for 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive memantine orally (PO) QD or twice daily (BID) for up to 24 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection and magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up every 2-3 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of small cell lung cancer within 5 years of registration. If the original histologic proof of malignancy is greater than 5 years, then pathological (i.e., more recent) confirmation is required (e.g., from a systemic or brain metastasis);

  * Patients with de novo or recurrent small cell lung cancer are permitted.
* Brain metastases =< 4 cm in largest diameter and outside a 5-mm margin around either hippocampus must be visible on contrast-enhanced magnetic resonance imaging (MRI) performed =< 21 days prior to study entry.

  * The total tumor volume must be 30 cm^3 or less. Lesion volume will be approximated by measuring the lesion's three perpendicular diameters on contrast enhanced, T1-weighted MRI and the product of those diameters will be divided by 2 to estimate the lesion volume (e.g. xyz/2). Alternatively, direct volumetric measurements via slice by slice contouring on a treatment planning software package can be used to calculate the total tumor volume.
  * Brain metastases can be diagnosed synchronous to the initial diagnosis of small cell lung cancer or metachronous to the initial diagnosis and management of small cell lung cancer.
  * Brain metastases must be diagnosed on MRI, which will include the following elements:

    * REQUIRED MRI ELEMENTS

      * Post gadolinium contrast-enhanced T1-weighted three-dimensional (3D) spoiled gradient (SPGR). Acceptable 3D SPGR sequences include magnetization prepared 3D gradient recalled echo (GRE) rapid gradient echo (MP-RAGE), turbo field echo (TFE) MRI, BRAVO (Brain Volume Imaging) or 3D Fast FE (field echo). The T1-weighted 3D scan should use the smallest possible axial slice thickness, not to exceed 1.5 mm.
      * Pre-contrast T1 weighted imaging (3D imaging sequence strongly encouraged).
      * A minimum of one axial T2 FLAIR (preferred) or T2 sequence is required. This can be acquired as a two dimensional (2D) or 3D image. If 2D, the images should be obtained in the axial plane.
    * ADDITIONAL RECOMMENDATIONS

      * Recommendation is that an axial T2 FLAIR (preferred) sequence be performed instead of a T2 sequence.
      * Recommendation is that that pre-contrast 3D T1 be performed with the same parameters as the post-contrast 3D T1.
      * Recommendation is that imaging be performed on a 3 Tesla (3T) MRI.
      * Recommendation is that the study participants be scanned on the same MRI instrument at each time point.
      * Recommendation is that if additional sequences are obtained, these should meet the criteria outlined in Kaufmann et al., 2020.
      * If additional sequences are obtained, total imaging time should not exceed 60 minutes.
      * If additional metastases not known at the time of registration/randomization or seen in the MRI used for eligibility are subsequently found on the radiation therapy (RT) planning MRI such that the total intacranial volume exceeds 30 cm^3, the patient is still considered eligible.
* History/physical examination
* Age >= 18
* Karnofsky performance status of >= 70
* Creatinine clearance >= 30 ml/min
* Following the diagnosis of brain metastases, patients can initiate and treat with systemic (chemotherapy and/or immunotherapy) before enrollment only if their brain metastases are asymptomatic and not located in eloquent locations (e.g., brainstem, pre-/post-central gyrus, visual cortex). However, within 21 days prior to enrollment, brain MRI must be repeated to confirm eligibility.

  * Patients with symptomatic brain metastases and/or brain metastases in eloquent locations (e.g., brainstem, pre-/post central gyrus, visual cortex) are eligible for enrollment on the trial; however, the specific treatment approach of starting with systemic therapy alone and delaying brain radiation is not recommended for these patients.
* Concurrent immunotherapy with brain radiation (SRS or HA-WBRT) is permitted.
* Negative urine or serum pregnancy test (in women of childbearing potential) within 14 days prior to registration. Women of childbearing potential and men who are sexually active must use contraception while on study.
* Patients may have had prior intracranial surgical resection.
* Because neurocognitive testing is the primary goal of this study, patients must be proficient in English or French Canadian.
* The patient must provide study-specific informed consent prior to study entry.

  * Patients with impaired decision-making capacity are not permitted on study.
* ELIGIBILITY CRITERIA PRIOR TO STEP 2 REGISTRATION
* The following baseline neurocognitive tests must be completed within 21 days prior to Step 2 registration: HVLT-R, TMT, and COWA. The neurocognitive test will be uploaded into RAVE for evaluation by Dr. Wefel. Once the upload is complete, within 3 business days a notification will be sent via email to the RA to proceed to Step 2.

  * NOTE: Completed baseline neurocognitive tests can be uploaded at the time of Step 1 registration.
* PRIOR TO STEP 2 REGISTRATION: The following baseline neurocognitive tests must be completed within 21 days prior to Step 2 registration: HVLT-R, TMT, and COWA. The neurocognitive tests will be uploaded into RAVE for evaluation by Dr. Wefel. Once the upload is complete, within 3 business days a notification will be sent via email to the RA to proceed to Step 2.

NOTE: Completed baseline neurocognitive tests can be uploaded at the time of Step 1 registration.

Exclusion Criteria:

* Planned infusion of cytotoxic chemotherapy on the same day as SRS or HA-WBRT treatment. Patients may have had prior chemotherapy. Concurrent immunotherapy is permitted.

  * For patients receiving fractionated SRS on an every-other-day basis, planned infusion of cytotoxic chemotherapy is not permitted between SRS treatments.
* Brainstem metastasis > 10 cm^3
* Prior allergic reaction to memantine.
* Patients with definitive leptomeningeal metastases.
* Known history of demyelinating disease such as multiple sclerosis.
* Contraindication to MR imaging such as implanted metal devices that are MRI-incompatible, allergy to MRI contrast that cannot be adequately addressed with pre-contrast medications, or foreign bodies that preclude MRI imaging. (Questions regarding MRI compatibility of implanted objects should be reviewed with the Radiology Department performing the MRI).
* Current use of (other N-methyl-D-aspartate [NMDA] antagonists) amantadine, ketamine, or dextromethorphan.
* Radiographic evidence of hydrocephalus or other architectural change of the ventricular system resulting in significant anatomic distortion of the hippocampus, including placement of external ventricular drain or ventriculoperitoneal shunt.

  * Mild cases of hydrocephalus not resulting in significant anatomic distortion of the hippocampus are permitted.
* Prior radiotherapy to the brain, including SRS, WBRT, or prophylactic cranial irradiation (PCI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to neurocognitive failure | Up to 1 year
  A failure is defined using the reliable change index (RCI) criteria, as measured by the Hopkins Verbal Learning Test - Revised (HVLT-R), Controlled Oral Word Association (COWA) test, and Trail Making Test (TMT) Parts A and B. The cumulative incidence approach will be used to estimate the percentage of failures while accounting for the competing risk of death.

SECONDARY OUTCOMES:
Preservation of neurocognitive function | 1 year
  Neurocognitive function will be measured by the HVLT-R, COWA, and TMT. The HVLT-R has 3 parts that will be analyzed separately: Total Recall, Delayed Recall, and Delayed Recognition. The TMT also has 2 parts that will be analyzed separately: TMT Part A and TMT Part B. The COWA has a single outcome measure that will be analyzed. Standardized scores that adjust for age, education, and sex when necessary will be analyzed.
Perceived difficulties in cognition | Up to 1 year
  Measured by Patient Reported Outcomes Measurement Information System (PROMIS). The total raw score for a PROMIS short form would be the sum of the values of the response to each question (therefore, for a short form which all questions are answered, the lowest possible score is 4 and the highest possible raw score is 20).
Symptom burden | Up to 1 year
  Measured by MD Anderson Symptom Inventory for brain tumor (MDASI-BT). Four subscales (symptom severity, symptom interference, neurologic factor, and cognitive factor score) as well as certain individual items (fatigue, neurologic factor items, and cognitive factor items) of the MDASI-BT will be analyzed.
Time to intracranial disease progression | From the date of randomization to the date of intracranial disease progression, assessed up to 10 years
  Time to any intracranial progression will be measured from the date of randomization to the date of intracranial disease progression. Death without an event will be treated as a competing risk. Alive patients without an event will be censored at their last known follow-up time. The percentage of patients with a failure will be determined using cumulative incidence.
Overall survival | From the date of randomization to the date of death, or otherwise, the last follow-up date on which the patient was reported alive, assessed up to 10 years
  Overall survival will be measured from the date of randomization to the date of death, or, otherwise, the last follow-up date on which the patient was reported alive. The Kaplan-Meier method (Kaplan 1958) will be used to calculate the percentage of patients alive.
Time to neurologic death | From the date of randomization to the date of neurologic death, assessed up to 10 years
  Time to neurologic death will be measured from the date of randomization to the date of neurologic death. Death without an event will be treated as a competing risk. Alive patients without an event will be censored at their last known follow-up time. The percentage of patients with a failure will be determined using cumulative incidence.
Salvage procedures used to manage recurrent intracranial disease | Up to 10 years
  Will be described by each arm.
Incidence of adverse events | Up to 10 years
  Graded by Common Terminology Criteria for Adverse Events version 5.0. Counts and frequencies will be provided for the worst grade AE experienced by the patient by treatment arm.
Development of cerebral necrosis | Up to 10 years

OTHER OUTCOMES:
Time to local brain recurrence (in brain lesions present at trial enrollment and treated with either stereotactic radiosurgery [SRS] or hippocampal-avoidant whole brain radiotherapy [HA-WBRT]) | Up to 10 years
Time to incidence of distant brain relapses | Up to 10 years
Time to leptomeningeal dissemination | Up to 10 years
White matter injury and hippocampal volume | 6 months
Time delay to salvage WBRT or HA-WBRT in patients on the SRS arm | Baseline to first salvage treatment, assessed up to 10 years
Cost and quality adjusted survival | Up to 1 year
  Measured using the European Quality of Life Five Dimension Five Level Scale Questionnaire.
Correlation between neurocognitive function and patient-reported outcomes | Up to 1 year
Estimates of treatment effect by sex | Up to 10 years
  Estimates of the primary outcome treatment effect and the corresponding 95% confidence intervals (CIs) by sex.
Estimates of treatment effect by race | Up to 10 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by race.
Estimates of treatment effect by ethnicity | Up to 10 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Vinai Gondi, Principal Investigator — NRG Oncology
Locations (224):
- United States (220):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Cherokee, Canton, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Rush-Copley Medical Center, Aurora, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Sands Cancer Center, Canandaigua, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Upstate Cancer Center Radiation Oncology at Oswego, Oswego, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Hill Radiation Oncology, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Saint Luke's Hospital-Quakertown Campus, Quakertown, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
- Canada (4):
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan